CLINICAL TRIAL: NCT06034860
Title: A Phase 1 Open-label, Multicenter, Dose-ranging Study to Investigate Safety and Tolerability, Efficacy, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of MT-8421 as Monotherapy and in Combination With Nivolumab in Patients With Selected Advanced Solid Cancer Types
Brief Title: Study of MT-8421 as Monotherapy and in Combination With Nivolumab in Patients With Selected Advanced Solid Cancer Types
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Termination
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-8421-001
Record Dates: First submitted 2023-08-23; First posted 2023-09-13 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Non Small Cell Lung Cancer; Hepatocellular Carcinoma; Melanoma; Renal Cell Carcinoma; Microsatellite Instability High; Mismatch Repair Deficiency; Mesothelioma; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Urothelial Carcinoma; Cervical Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Renal Cell; Turcot syndrome; Mesothelioma; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Uterine Cervical Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A- Dose Escalation Monotherapy (Experimental): Part A- Dose escalation of MT-8421 monotherapy in patients with selected advanced solid tumors.
  The assigned dose level of MT-8421 will be given as an intravenous (IV) infusion over about 30 minutes on the same day every week (i.e. on day 1, day 8, day 15, and day 22 of each 28-day cycle).
  Interventions: Drug: MT-8421
- Part A- Dose Escalation Combination Therapy (Experimental): Part A- Dose escalation of MT-8421 in combination with nivolumab in patients with selected advanced solid tumors.
  The assigned dose level of MT-8421 will be given as an intravenous (IV) infusion over about 30 minutes prior to the infusion of 480 mg nivolumab. MT-8421 will be given on the same day every week (i.e. on day 1, day 8, day 15, and day 22 of each 28-day cycle). Nivolumab will be given on the first day of each cycle beginning at cycle 2.
  Interventions: Drug: MT-8421; Drug: Nivolumab
- Part B Dose Expansion Monotherapy (Experimental): Part B- Dose expansion of MT-8421 monotherapy in patients with selected advanced solid tumors.
  Part B monotherapy will include two expansion groups: Group B1 (NSCLC) and group B2 (HCC).
  The assigned dose level of MT-8421 determined in Part A will be given as an intravenous (IV) infusion over about 30 minutes on the same day every week (i.e. on day 1, day 8, day 15, and day 22 of each 28-day cycle).
  Interventions: Drug: MT-8421
- Part B Dose Expansion Combination (Experimental): Part B- Dose escalation of MT-8421 in combination with nivolumab in patients with selected advanced solid tumors.
  Part B combination therapy will include two expansion groups: Group B3 (Melanoma) and Group B4 (RCC).
  The assigned dose level of MT-8421 determined in Part A will be given as an intravenous (IV) infusion over about 30 minutes prior to the infusion of 480 mg nivolumab. MT-8421 will be given on the same day every week (i.e. on day 1, day 8, day 15, and day 22 of each 28-day cycle). Nivolumab will be given on the first day of each cycle beginning at cycle 2.
  Interventions: Drug: MT-8421; Drug: Nivolumab

INTERVENTIONS:
Drug: MT-8421 — Experimental treatment with MT-8421
Drug: Nivolumab — 480 mg nivolumab administered on Day 1 of each cycle starting with Cycle 2 for all combination dose escalation and dose expansion cohorts
  Arms: Part A- Dose Escalation Combination Therapy; Part B Dose Expansion Combination

SUMMARY:
This is a Phase 1, open-label, dose escalation and expansion study of MT-8421 (an Engineered Toxin Body (ETB)) as monotherapy and in combination with nivolumab in patients with selected advanced solid cancer types. MT-8421 is an investigational drug that specifically targets and depletes cytotoxic T-lymphocytes-associated protein 4 (CTLA-4) expressing cells in an effort to directly dismantle the tumor microenvironment for the treatment of patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is conducted in two parts. The study will enroll up to 200 total participants (up to 40 in Part A and up to 160 in Part B).

Part A (Dose Escalation) is designed to estimate the maximum tolerated dose (MTD) of MT-8421 as monotherapy and in combination with nivolumab.

Part B (Dose Expansion) is designed to identify the dose(s) to be studied in Phase 2.

The drug being tested in this study is called MT-8421. The study will evaluate safety, tolerability, efficacy, pharmacokinetics, pharmacodynamics, and immunogenicity of MT-8421 as monotherapy and in combination with nivolumab in patients with selected advanced solid cancer types.

MT-8421 will be given as an intravenous (IV) infusion on Days 1, 8, 15, and 22 of a 28-day cycle. H1 and H2 blockers and anti-pyretics will be given to all patients as pre-medication prior to each dose in Cycle 1. Anti-pyretics will be required for 24 hours after the first dose in Cycle 1. Use of pre-medication will be at the discretion of the Investigator for subsequent doses.

In Parts A and B, a subject may participate for the following three (3) periods:

* Screening Period- up to 28 days before the first dose of MT-8421
* Treatment Period- active period where a subject will receive doses of MT-8421 over a 28-day treatment period.
* Follow-up Period- up to 24 months after the second short term follow up visit.

In both parts of the study, participants can receive MT-8421 until their cancer worsens, side effects prevent further study treatment, or until the participant leaves the study for other reasons decided by the participant, the study doctor, or the sponsor of the study. After the second short term follow up visit participants will have a check -up of their disease every 12 weeks for 24 months.

The overall duration of the study will vary for each participant because study treatment will continue until unacceptable toxicity, withdrawal of consent, death, termination of the study by the sponsor, or fulfilment of another discontinuation criterion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable, locally advanced, or metastatic melanoma, HCC, NSCLC, RCC, MSI-H/dMMR malignancies, urothelial carcinoma, esophageal squamous cell carcinoma, mesothelioma, SCCHN, or cervical carcinoma not amenable to standard treatment, or standard treatment is not available, or in the Investigator's opinion, the standard treatment would not be in the patient's best interest.

Part A only: Evaluable only or measurable disease according to RECIST v1.1 Part B only: At least 1 measurable tumor lesion according to RECIST v1.1

* Prior treatment must include a PD-1 or programmed cell death - ligand 1 (PD-L1) inhibitor. Prior treatment with a CTLA-4 inhibitor is not required.
* Eastern Cooperate Oncology Group (ECOG) performance score of 0 or 1
* Adequate bone marrow function, as determined by:

  * Absolute neutrophil count (ANC) ≥ 1500/ μL (should not have received growth factors within 2 weeks prior to screening)
  * Platelet count ≥ 75,000/ μL
  * Hemoglobin ≥ 8.0 g/dL (no red blood cell transfusion within 2 weeks of study treatment start is allowed)
* Adequate renal function, based on estimated creatinine clearance (eCrCl) ≥ 50 mL/min, calculated by the Cockcroft-Gault equation.
* Adequate hepatic function, as determined by:

  * Total bilirubin ≤ 1.5x upper limit of normal (ULN) or ≤ 2x ULN direct bilirubin for patients with Gilbert's Syndrome
  * Aspartate transaminase (AST) ≤ 3x ULN (or ≤ 5x ULN if liver metastasis or HCC).
  * Alanine transaminase (ALT) ≤ 3x ULN (or ≤ 5x ULN if liver metastasis or HCC).
  * Adequate serum albumin (albumin ≥ 2.5 g/dL)
* Availability of a lesion that can be biopsied with acceptable risk.
* Patients capable of bearing children must have a negative highly sensitive pregnancy test within 72 hours before the start of treatment. Patients who are postmenopausal (> 1 year since last menstrual cycle) or permanently sterilized (e.g., bilateral tubal occlusion, hysterectomy, bilateral salpingectomy) may be considered as not of reproductive potential.
* Patients of reproductive potential must agree either to abstain continuously from heterosexual intercourse or to use a highly effective birth control method from signing the informed consent form (ICF) until 30 days after the last dose of MT-8421 and/or 5 months after the last dose of nivolumab for patients capable of bearing children and until 90 days after the last dose of MT-8421 for patients capable of fathering a child. Patients must not donate sperm during the study and for 90 days after the last dose of nivolumab or MT-8421.

Exclusion Criteria:

* Unwilling or unable to undergo 2 sets of 3 to 6 core tumor biopsies: one set at study baseline (prior to first dose of study drug) and one set between Weeks 6 through 8. A final optional set will be collected time of disease progression.
* Received approved or investigational treatment for the disease under study (except ipilimumab) where Exclusion Criterion 4 applies, requiring a washout that will be dependent upon prior ipilimumab dose and planned MT-8421 dose) within 4 weeks before the start of treatment. For small molecules [Molecular Weight (MW) < 0.9 kDa], the washout is 5 half-lives, but at least 2 weeks.
* Received tremelimumab within 30 days or ipilimumab 3 mg/kg within 60 days or ipilimumab 1 mg/kg within 30 days before the start of treatment. Once dose cohort of 32 µg/kg MT-8421 has been completed in dose escalation, a 30-day washout of ipilimumab is acceptable irrespective of prior dose.
* Any concurrent cancer treatment, apart from local treatment of non-target lesions for palliative intent (e.g., local surgery or radiotherapy). Patient must have recovered from the effects of the local treatment and be discussed with the medical monitor.
* History or current evidence of another neoplastic disease, except cervical carcinoma in situ; superficial non-invasive bladder tumors, curatively treated; Stage I to II non-melanoma skin cancer; prostate cancer managed by active surveillance; or any previous cancer curatively treated < 2 years before the start of treatment.
* Active autoimmune disease that required systemic treatment in the past. Patients who have not required systemic treatment for at least 2 years may be enrolled if permission is provided after discussion with the Medical Monitor (replacement therapy, e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is allowed)
* Evidence of active, non-infectious ≥ Grade 2 pneumonitis or current evidence of ≥ Grade 3 other underlying pulmonary disease.
* Ongoing > Grade 1 immune-related toxicity caused by prior CPI therapy (i.e., PD-1 inhibitors, PDL1 inhibitors, or CTLA-4 inhibitors). Patients with stable endocrinological AEs (e.g., hypothyroidism, adrenal insufficiency, hypopituitarism, or diabetes mellitus) must have been on a stable dose of supplemental therapy for at least 2 weeks before screening to be eligible for this study. History of repeat Grade 2 pneumonitis or myocarditis on previous CPI and/or Grade 3 irAE on previous CPI treatment.
* Current evidence of new or growing central nervous system (CNS) metastases during screening. Patients with known CNS metastases will be eligible if they meet all the following criteria:

  * Received radiotherapy or another appropriate therapy for the CNS metastases, if clinically Indicated
  * Have stable CNS disease on the computed tomography (CT) or magnetic resonance imaging (MRI) scan within 4 weeks before signing the ICF compared with prior neuroimaging.
* History or current evidence of significant cardiovascular disease before the start of treatment.
* Current evidence of active, uncontrolled hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV) (evidenced by detectable viral load by polymerase chain reaction) or acquired immunodeficiency syndrome (AIDS)-related illness.

  * Serology and virology measurements are not required to be performed at screening, but any previously reported results should be used for eligibility purposes. Investigators will test per their discretion
  * Patients with a history of treated hepatitis C and non-quantifiable hepatitis C virus- ribonucleic acid (RNA) may be enrolled.
  * Patients on treatment for hepatitis B, hepatitis C, and/or HIV will be eligible if they have undetectable viral load (patients with HIV with CD4+ T-cell [CD4+] counts ≥ 350 cells/µL may be enrolled).
* Patients with unintentional weight loss greater than 10% of their body weight over the preceding 2 months or less prior to first dose in the first cycle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 28 day cycle
  Evaluation of safety and tolerability of MT-8421 as measured by number of participants with Adverse Events, dose limiting toxicities (DLTs), abnormal physical exam findings, abnormal laboratory test results, abnormal radiographic findings, and/or patient reported symptoms
To confirm the recommended Phase 2 dose (RP2D) of MT-8421 as monotherapy and in combination with nivolumab in patients with selected advanced solid tumor types. | 28 day cycle
  Incidence of AEs
Proportion of participants with objective response | Up to two years (Part B)
  Objective response rate (ORR) defined as the proportion of participants with either a complete response or a partial response as determined by investigator assessment using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Objective response rate to assess preliminary efficacy | Up to two years (Parts A)
  Objective response rate (ORR) defined as the proportion of participants with either a complete response or a partial response as determined by investigator assessment using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Duration of response to assess preliminary efficacy | Up to two years (Parts A)
  Duration of response defined for participants with confirmed complete response or partial response as the time from the first documented tumor response to the date of radiographic progression progressive disease per RECIST v1.1
Time to response to assess preliminary efficacy | Up to two years (Parts A)
  Time to response defined as the time from the date of the first dose of the study treatment to the date of the first documentation of response (partial response or better) per RECIST v1.1
Progression-free survival to assess preliminary efficacy | Up to two years (Parts A)
  Progression free survival defined as the time from the start of treatment with MT-8421 to the date of radiographic progressive disease per RECIST v1.1 or death from any cause, not including clinical progression
Disease control rate to assess preliminary efficacy | Up to two years (Parts A)
  Disease control rate defined as proportion of patients who have achieved complete response, partial response and stable disease
Characterize the pharmacokinetic (PK) profile of MT-8421 given as monotherapy and in combination with nivolumab in patients with selected advanced solid tumor types | Up to two years (Parts A)
  Maximum observed plasma concentration (Cmax)
Characterize the pharmacokinetic (PK) profile of MT-8421 given as monotherapy and in combination with nivolumab in patients with selected advanced solid tumor types | Up to two years (Parts A and B)
  Half-life (t1/2)
Characterize the pharmacokinetic (PK) profile of MT-8421 given as monotherapy and in combination with nivolumab in patients with selected advanced solid tumor types | Up to two years (Parts A and B)
  Area under the concentration-time curve (AUC) from time zero to the last measurable concentration (AUC0-t), total exposure (AUC0-∞)
Characterize the pharmacokinetic (PK) profile of MT-8421 given as monotherapy and in combination with nivolumab in patients with selected advanced solid tumor types | Up to two years (Parts A and B)
  Clearance (CL)
Characterize the pharmacokinetic (PK) profile of MT-8421 given as monotherapy and in combination with nivolumab in patients with selected advanced solid tumor types | Up to two years (Parts A and B)
  Volume of distribution at steady-state (Vss)
Evaluate the immunogenicity of MT-8421 in patients with selected advanced solid tumors. | Up to two years (Parts A and B)
  Anti-drug antibodies (ADA), Neutralizing antibodies (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: Admasu Mamuye, MD, Study Director — Molecular Templates
Locations (5):
- United States (5):
  - The Angeles Clinic, Los Angeles, California
  - Horizon Oncology Research, LLC, Lafayette, Indiana
  - Washington University in St. Louis, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - NEXT Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No